CLINICAL TRIAL: NCT05957848
Title: Guanfacine Extended-release Randomised Controlled Trial for Adolescents With Cannabis usE (GRACE)
Brief Title: Guanfacine Extended-release for Adolescents With Cannabis Use
Acronym: GRACE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Orygen (Other)
Collaborators: Youth Support and Advocacy Service (Unknown); University of Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22389
Record Dates: First submitted 2023-06-15; First posted 2023-07-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Guanfacine; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guanfacine extended-release (Experimental): Guanfacine extended-release (target dose 4 mg), once daily for approximately 12 weeks plus treatment as usual
  Interventions: Drug: Guanfacine Extended Release Oral Tablet; Behavioral: Residential withdrawal; Behavioral: Engagement with alcohol and other drug services
- Placebo (Placebo Comparator): Placebo once daily for approximately 12 weeks plus treatment as usual
  Interventions: Behavioral: Residential withdrawal; Behavioral: Engagement with alcohol and other drug services; Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine Extended Release Oral Tablet — Target dose 4 mg daily
  Other Names: Intuniv; Guanfacine XR
  Arms: Guanfacine extended-release
Behavioral: Residential withdrawal — 4-14 days in residential withdrawal treatment
Behavioral: Engagement with alcohol and other drug services — Ongoing engagement with a youth drug and alcohol service for counselling or other support for the duration of the study
Drug: Placebo — Placebo capsule taken daily
  Arms: Placebo

SUMMARY:
A randomized controlled trial to assess the efficacy of extended-release guanfacine to reduce cannabis use frequency in young people with cannabis use disorder following a period of monitored abstinence.

ELIGIBILITY:
Inclusion Criteria:

1. 12-25 years of age (inclusive) at consent;
2. Seeking treatment for cannabis use;
3. DSM-5 Cannabis Use Disorder, mild, moderate or severe;
4. Self-reported cannabis use on average at least 5 days/week during the 28 days prior to screening with a THC positive urine drug screen on the day of screening; and
5. Able to provide informed consent (both adequate IQ and English fluency; <18-year-olds will provide consent themselves in addition to parent/guardian consent).

Exclusion Criteria:

1. DSM-5 substance use disorder (moderate or severe) except cannabis or nicotine;
2. Any unstable medical, psychiatric or neurological condition or medical contraindicating study participation;
3. Diagnosis of a psychotic or bipolar illness;
4. Acute suicidality as assessed by clinician;
5. Prescribed antipsychotics, benzodiazepines or other sedative medications, or other medications for the treatment of ADHD. If prescribed antidepressants, the participant must have been on a stable dose for more than 2 weeks at screening;
6. A history of heart disease or cardiac risk factors (e.g. arrhythmias);
7. Abnormal liver or thyroid function as indicated by clinically-significant findings on blood tests;
8. Pregnancy, breast feeding or, if sexually active and able to become pregnant, no effective contraception.
9. Intention to enter residential rehabilitation after treatment in the YSAS residential withdrawal facility.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy - change from baseline in cannabis use frequency following monitored abstinence | Baseline and weekly in the 4 week outpatient phase immediately following discharge from residential withdrawal
  Change from baseline in average frequency of cannabis use (days of use/week) in the 4 weeks immediately following discharge from residential withdrawal, assessed weekly using the Timeline Follow-Back.

SECONDARY OUTCOMES:
Change from baseline in cannabis use frequency following monitored abstinence (categorical) | Baseline and weekly in the 4 weeks immediately following discharge from residential withdrawal
  Change from baseline in average frequency of cannabis use in the 4 weeks immediately following discharge from residential withdrawal, assessed weekly using the Timeline Follow-Back and categorized as follows: heavy use (5-7 days per week), moderate use (3-5 days) or light use (0-1 days)
Cannabis exposure | Approximately weekly between Baseline (week 0) and the end of treatment visit (week C7), approximately 12 weeks from baseline
  The number of urine toxicology tests that are positive for cannabis exposure
Change from baseline in cannabis use disorder symptoms | Baseline and end of Maintenance phase (4 weeks post discharge from residential withdrawal)
  Change from baseline in number of cannabis use disorder symptoms endorsed at end of treatment as indexed by the Structured Clinical Interview for DSM-5 (SCID-5)
Cannabis withdrawal symptoms during residential withdrawal admission | Daily during residential treatment for 4 to 14 days
  Measured with the Cannabis Withdrawal Scale
Sleep quality (subjective) during residential withdrawal admission | Daily during residential treatment for 4 to 14 days
  Measured with the PROMIS Sleep Disturbance Scale
Cannabis craving during residential withdrawal admission | Daily during residential treatment for 4 to 14 days
  Measured with the Brief Substance Craving Scale - Cannabis
Sleep quality (objective) during residential withdrawal admission | Daily during residential treatment for 4 to 14 days
  Measured with wrist actigraphy
Food intake during residential withdrawal admission | Daily during residential treatment for 4 to 14 days
  Measured with a food intake dairy
Treatment engagement (residential) | Baseline to end of treatment
  Measured as the longest consecutive length of stay in residential withdrawal (4-14 days)
Treatment engagement (outpatient) | Baseline to end of treatment
  Measured as the number of outpatient alcohol and other drug counselling sessions completed
Change from baseline in daily functioning - social and occupational | Baseline and end of maintenance period assessments (4 weeks post discharge from residential withdrawal)
  Measured with the Social and Occupational Functioning Assessment scale (SOFAS)
Change from baseline in daily functioning - multidimensional | Baseline and end of maintenance period assessments (4 weeks post discharge from residential withdrawal)
  Measured with the Multidimensional Adolescent Functioning Scale (MAFS)
Change from baseline in daily functioning - social inclusion | Baseline and end of maintenance period assessments (4 weeks post discharge from residential withdrawal)
  Measured with the Filia Social Inclusion Measure - 16 item scale (FSIM-16).

CONTACTS AND LOCATIONS:
Locations (1):
- Orygen, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No